CLINICAL TRIAL: NCT04761523
Title: The Effect of Dietary Fat Content on the Recurrence of Pancreatitis (EFFORT): Protocol of a Multicentre Randomized Controlled Trial
Brief Title: The Effect of Dietary Fat Content on the Recurrence of Pancreatitis
Acronym: EFFORT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pecs (Other)
Responsible Party: Principal Investigator, Dr Hegyi Péter, Principal Investigator, Director of the Centre for Translational Medicine at University of Pécs, University of Pecs
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 40304-11/2020/EÜIG
Record Dates: First submitted 2021-02-15; First posted 2021-02-21 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Acute Pancreatitis
Keywords: acute pancreatitis; dietary fat; low-fat diet; pancreatitis recurrence
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Doctors caring for the participants and assessors of all other outcomes (laboratory parameters, BMI, blood pressure, adverse events) as well as statisticians handling the data will be blinded to the participants' allocated group. Outcome assessors will be not avare of the allocated interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reduced fat arm (Active Comparator): Daily calorie intake will be composed of 15% fat, 65% carbohydrates, 20% proteins
  Interventions: Behavioral: Dietary intervention: reduced fat diet
- Standard healthy diet arm (Active Comparator): Daily calorie intake will be composed of 30% fat, 50% carbohydrates and 20% proteins.
  Interventions: Behavioral: Dietary intervention: standard healthy diet

INTERVENTIONS:
Behavioral: Dietary intervention: reduced fat diet — Participants will receive a dietary intervention, and will be proposed to adhere to a diet with a 15% fat, 65% carbohydrate, 20% protein content.
  Arms: Reduced fat arm
Behavioral: Dietary intervention: standard healthy diet — Participants will receive a dietary intervention, and will be proposed to adhere to a diet with a 30% fat, 50% carbohydrate, 20% protein content.
  Arms: Standard healthy diet arm

SUMMARY:
This trial aims to test the effects of two different diets on the recurrence of acute pancreatitis, and acute pancreatitis associated mortality.

DETAILED DESCRIPTION:
Around 20% of patients with acute pancreatitis (AP) will go on to have acute recurrent pancreatitis (ARP) and 10% progress to chronic pancreatitis (CP). While interventions to avoid recurrences exist for the two most common causes - removal of the cholecyst in the case of biliary, and alcohol seccation in the case of alcoholic - a method to prevent idiopathic pancreatitis is not yet known. Although none of the guidelines suggest the administration of low fat diet, it is recommended by physicians to all pancreatitis patients are. Our aim is to conduct a randomized controlled trial, to assess the problem of dietary fat reduction on the recurrence of acute pancreatitis Patients, who had at least two acute pancreatitis episodes in the preceding 2 year will be approached to participate in the study and to either to be randomized to the 'reduced fat diet' (15% fat, 65% carbohydrate, 20% protein) or to the 'standard healthy diet' (30% fat, 50% carbohydrate, 20% protein; based on WHO recommendations) group. During the 2 year long followup, participants will receive repeated dietary intervention at 3, 6, 12, 18, 24 months, they will completer food frequency questionnaires and their data regarding mortality, BMI, cardiovascular parameters and serum lipid values will be recorded The EFFORT trial will determine the effect of modified dietary fat content on the recurrence of AP, mortality, serum lipids and weight loss in idiopathic cases.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with at least two episodes of acute pancreatitis in the 2 years preceding the inclusion with
* The last episode being idiopathic, who are
* Older than 14 years.

Exclusion Criteria:

* Individuals already receiving regular nutritional guidance (with medical indication),
* Individuals in critical condition or in terminal stage of cancer (with an expected survival <2 years) ,
* Individuals undergoing treatment for active malignancy,
* Individuals with uncontrolled diabetes mellitus (admitted lack of compliance with antidiabetic therapy / HbA1c >6.5% / indication of uncontrolled diabetes mellitus in last 24 months' anamnesis / newly discovered diabetes mellitus)
* Individuals with known cholecystolithiasis
* Individuals who are pregnant or nursing
* Individuals with a BMI < 18.5
* Individuals who are regularly receiving systemic corticosteroids
* Individuals consuming more alcohol than: 5 units per day or 15 units per week for men; 4 units per day or 8 units per week for women.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 384 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of recurrent acute pancreatitis and/or all-cause mortality | Data will be recorded during the 3-6-12-18-24 months followup visits
  The recurrence of acute pancreatitis (given as a rate of event) AND/OR all-cause mortality.

SECONDARY OUTCOMES:
Proportion of pancreas specific mortality | Data will be recorded during the 3-6-12-18-24 months followup visits
  Mortality of a pancreatic cause
Proportion of cardiosvascular cause mortality | Data will be recorded during the 3-6-12-18-24 months followup visits
  Mortality of a cardiovascular cause.
Proportion of newly diagnosed chronic pancreatitis patients | Data will be recorded during the 3-6-12-18-24 months followup visits
  Newly diagnosed chronic pancreatitis.
Changes in BMI | Data will be recorded az baseline, and during the 3-6-12-18-24 months followup visits
  Changes in BMI compared to baseline both in total and percentage
Serum total cholesterol | Data will be recorded during the 3-6-12-18-24 months followup visits
  Serum total cholesterol absolute value
Change in serum total cholesterol | Data will be recorded at baseline, and during the 3-6-12-18-24 months followup visits
  Serum total cholesterol compared to baseline
Serum triglyceride | Data will be recorded during the 3-6-12-18-24 months followup visits
  Serum triglyceride absolute value
Change in serum triglyceride | Data will be recorded at baseline, and during the 3-6-12-18-24 months followup visits
  Serum triglyceride compared to baseline
Serum high density liporpotein(HDL)-cholesterol | Data will be recorded during the 3-6-12-18-24 months followup visits
  Serum high density liporpotein(HDL)-cholesterol absolute value
Change in serum high density liporpotein(HDL)-cholesterol | Data will be recorded at baseline, and during the 3-6-12-18-24 months followup visits
  Serum high density liporpotein(HDL)-cholesterol compared to baseline
Serum low density liporpotein(LDL)-cholesterol | Data will be recorded during the 3-6-12-18-24 months followup visits
  Serum low density liporpotein(LDL)-cholesterol absolute value
Change in serum low density liporpotein(LDL)-cholesterol | Data will be recorded at baseline, and during the 3-6-12-18-24 months followup visits
  Serum low density liporpotein(LDL)-cholesterol compared to baseline
Systolic blood pressure value | Data will be recorded during the 3-6-12-18-24 months followup visits
  Systolic blood pressure absolute value
Change in systolic blood pressure | Data will be recorded az baseline, and during the 3-6-12-18-24 months followup visits
  Systolic blood pressure compared to baseline
Diastolic blood pressure | Data will be recorded during the 3-6-12-18-24 months followup visits
  Diastolic blood pressure absolute value
Change in siastolic blood pressure | Data will be recorded at baseline, and during the 3-6-12-18-24 months followup visits
  Diastolic blood pressure compared to baseline
Adherence to dietary recommendations as determined by the result of the food frequency questionnaire | Data will be recorded during the 3-6-12-18-24 months followup visits
  Adherence to dietary recommendations as determined by the result of the food frequency questionnaire
Adverse effects | Data will be recorded during the 3-6-12-18-24 months followup visits
  Adverse effects given as rate of events
Serum albumin value | Data will be recorded during the 3-6-12-18-24 months followup visits
  Serum albumin absolute value
Change in serum albumin value | Data will be recorded at baseline, and during the 3-6-12-18-24 months followup visits
  Serum albumin value compared to baseline
Proportion of current smokers | Data will be recorded at baseline, and during the 3-6-12-18-24 months followup visits
  Current smoking at each visit
Quality of life questionnaire on mobility, self-care, usual activities, pain/discomfort and anxiety/depression | Data will be recorded at baseline, and during the 3-6-12-18-24 months followup visits
  Quality of life assessed by the EQ-5D-5L questionnaire
Muscle strength | Data will be recorded at baseline, and during the 3-6-12-18-24 months followup visits
  Muscle strength using a handgrip dynamometer
Vitamin A value | Data will be recorded at baseline, and during the 3-6-12-18-24 months followup visits
  Vitamin A absolute value
Change in vitamin A value | Data will be recorded at baseline, and during the 3-6-12-18-24 months followup visits
  Change in vitamin A value compared to baseline
Vitamin D value | Data will be recorded at baseline, and during the 3-6-12-18-24 months followup visits
  Vitamin D absolute value
Change in vitamin D value | Data will be recorded at baseline, and during the 3-6-12-18-24 months followup visits
  Change in vitamin D value compared to baseline
Vitamin E value | Data will be recorded at baseline, and during the 3-6-12-18-24 months followup visits
  Vitamin E absolute value
Change in vitamin E value | Data will be recorded at baseline, and during the 3-6-12-18-24 months followup visits
  Change in vitamin E value compared to baseline
Vitamin K value | Data will be recorded at baseline, and during the 3-6-12-18-24 months followup visits
  Vitamin K absolute value
Change in vitamin K value | Data will be recorded at baseline, and during the 3-6-12-18-24 months followup visits
  Change in vitamin K value compared to baseline
Change in smoking | Data will be recorded at baseline, and during the 3-6-12-18-24 months followup visits
  Change in smoking compared to baseline
Change in quality of life | Data will be recorded at baseline, and during the 3-6-12-18-24 months followup visits
  Change in quality of life assessed by the EQ-5D-5L questionnaire compared to baseline
Change in muscle strength | Data will be recorded at baseline, and during the 3-6-12-18-24 months followup visits
  Change in muscle strength using a handgrip dynamometer compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Péter Hegyi, MD, PhD, DSc, Study Chair — Insitute for Translational Medicine, University of Pécs, Medical School, Pécs, Hungary
Locations (1):
- Division of Pancreatic Diseases, Heart and Vascular Center, Semmelweis University, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spanier BW, Dijkgraaf MG, Bruno MJ. Epidemiology, aetiology and outcome of acute and chronic pancreatitis: An update. Best Pract Res Clin Gastroenterol. 2008;22(1):45-63. doi: 10.1016/j.bpg.2007.10.007. PMID 18206812
- [Background] Sankaran SJ, Xiao AY, Wu LM, Windsor JA, Forsmark CE, Petrov MS. Frequency of progression from acute to chronic pancreatitis and risk factors: a meta-analysis. Gastroenterology. 2015 Nov;149(6):1490-1500.e1. doi: 10.1053/j.gastro.2015.07.066. Epub 2015 Aug 20. PMID 26299411
- [Background] Working Group IAP/APA Acute Pancreatitis Guidelines. IAP/APA evidence-based guidelines for the management of acute pancreatitis. Pancreatology. 2013 Jul-Aug;13(4 Suppl 2):e1-15. doi: 10.1016/j.pan.2013.07.063. PMID 24054878
- [Background] Tenner S, Baillie J, DeWitt J, Vege SS; American College of Gastroenterology. American College of Gastroenterology guideline: management of acute pancreatitis. Am J Gastroenterol. 2013 Sep;108(9):1400-15; 1416. doi: 10.1038/ajg.2013.218. Epub 2013 Jul 30. PMID 23896955
- [Background] Crockett SD, Wani S, Gardner TB, Falck-Ytter Y, Barkun AN; American Gastroenterological Association Institute Clinical Guidelines Committee. American Gastroenterological Association Institute Guideline on Initial Management of Acute Pancreatitis. Gastroenterology. 2018 Mar;154(4):1096-1101. doi: 10.1053/j.gastro.2018.01.032. Epub 2018 Feb 3. No abstract available. PMID 29409760
- [Background] Prizment AE, Jensen EH, Hopper AM, Virnig BA, Anderson KE. Risk factors for pancreatitis in older women: the Iowa Women's Health Study. Ann Epidemiol. 2015 Jul;25(7):544-8. doi: 10.1016/j.annepidem.2014.12.010. Epub 2015 Jan 7. PMID 25656921
- [Background] Setiawan VW, Pandol SJ, Porcel J, Wei PC, Wilkens LR, Le Marchand L, Pike MC, Monroe KR. Dietary Factors Reduce Risk of Acute Pancreatitis in a Large Multiethnic Cohort. Clin Gastroenterol Hepatol. 2017 Feb;15(2):257-265.e3. doi: 10.1016/j.cgh.2016.08.038. Epub 2016 Sep 5. PMID 27609706
- [Background] Oskarsson V, Sadr-Azodi O, Discacciati A, Orsini N, Wolk A. Overall diet quality and risk of recurrence and progression of non-gallstone-related acute pancreatitis: a prospective cohort study. Eur J Nutr. 2018 Oct;57(7):2537-2545. doi: 10.1007/s00394-017-1526-8. Epub 2017 Aug 30. PMID 28856418
- [Background] Cuevas A, Miquel JF, Reyes MS, Zanlungo S, Nervi F. Diet as a risk factor for cholesterol gallstone disease. J Am Coll Nutr. 2004 Jun;23(3):187-96. doi: 10.1080/07315724.2004.10719360. PMID 15190042
- [Background] Thomas T, Mah L, Barreto SG. Systematic review of diet in the pathogenesis of acute pancreatitis: a tale of too much or too little? Saudi J Gastroenterol. 2012 Sep-Oct;18(5):310-5. doi: 10.4103/1319-3767.101124. PMID 23006458
- [Background] Lindkvist B, Appelros S, Regner S, Manjer J. A prospective cohort study on risk of acute pancreatitis related to serum triglycerides, cholesterol and fasting glucose. Pancreatology. 2012 Jul-Aug;12(4):317-24. doi: 10.1016/j.pan.2012.05.002. Epub 2012 May 10. PMID 22898632
- [Background] Cappell MS. Acute pancreatitis: etiology, clinical presentation, diagnosis, and therapy. Med Clin North Am. 2008 Jul;92(4):889-923, ix-x. doi: 10.1016/j.mcna.2008.04.013. PMID 18570947
- [Background] Biczo G, Vegh ET, Shalbueva N, Mareninova OA, Elperin J, Lotshaw E, Gretler S, Lugea A, Malla SR, Dawson D, Ruchala P, Whitelegge J, French SW, Wen L, Husain SZ, Gorelick FS, Hegyi P, Rakonczay Z Jr, Gukovsky I, Gukovskaya AS. Mitochondrial Dysfunction, Through Impaired Autophagy, Leads to Endoplasmic Reticulum Stress, Deregulated Lipid Metabolism, and Pancreatitis in Animal Models. Gastroenterology. 2018 Feb;154(3):689-703. doi: 10.1053/j.gastro.2017.10.012. Epub 2017 Oct 23. PMID 29074451
- [Background] Zhang X, Cui Y, Fang L, Li F. Chronic high-fat diets induce oxide injuries and fibrogenesis of pancreatic cells in rats. Pancreas. 2008 Oct;37(3):e31-8. doi: 10.1097/MPA.0b013e3181744b50. PMID 18815536
- [Background] Czako L, Szabolcs A, Vajda A, Csati S, Venglovecz V, Rakonczay Z Jr, Hegyi P, Tiszlavicz L, Csont T, Posa A, Berko A, Varga C, Varga Ilona S, Boros I, Lonovics J. Hyperlipidemia induced by a cholesterol-rich diet aggravates necrotizing pancreatitis in rats. Eur J Pharmacol. 2007 Oct 15;572(1):74-81. doi: 10.1016/j.ejphar.2007.05.064. Epub 2007 Jun 13. PMID 17628538
- [Background] Nordback I, Pelli H, Lappalainen-Lehto R, Jarvinen S, Raty S, Sand J. The recurrence of acute alcohol-associated pancreatitis can be reduced: a randomized controlled trial. Gastroenterology. 2009 Mar;136(3):848-55. doi: 10.1053/j.gastro.2008.11.044. Epub 2008 Nov 27. PMID 19162029
- [Background] Bueno NB, de Melo IS, de Oliveira SL, da Rocha Ataide T. Very-low-carbohydrate ketogenic diet v. low-fat diet for long-term weight loss: a meta-analysis of randomised controlled trials. Br J Nutr. 2013 Oct;110(7):1178-87. doi: 10.1017/S0007114513000548. Epub 2013 May 7. PMID 23651522
- [Background] Mansoor N, Vinknes KJ, Veierod MB, Retterstol K. Effects of low-carbohydrate diets v. low-fat diets on body weight and cardiovascular risk factors: a meta-analysis of randomised controlled trials. Br J Nutr. 2016 Feb 14;115(3):466-79. doi: 10.1017/S0007114515004699. PMID 26768850
- [Background] Lu M, Wan Y, Yang B, Huggins CE, Li D. Effects of low-fat compared with high-fat diet on cardiometabolic indicators in people with overweight and obesity without overt metabolic disturbance: a systematic review and meta-analysis of randomised controlled trials. Br J Nutr. 2018 Jan;119(1):96-108. doi: 10.1017/S0007114517002902. Epub 2017 Dec 7. PMID 29212558
- [Background] Nordmann AJ, Nordmann A, Briel M, Keller U, Yancy WS Jr, Brehm BJ, Bucher HC. Effects of low-carbohydrate vs low-fat diets on weight loss and cardiovascular risk factors: a meta-analysis of randomized controlled trials. Arch Intern Med. 2006 Feb 13;166(3):285-93. doi: 10.1001/archinte.166.3.285. PMID 16476868
- [Background] Marta K, Szabo AN, Pecsi D, Varju P, Bajor J, Godi S, Sarlos P, Miko A, Szemes K, Papp M, Tornai T, Vincze A, Marton Z, Vincze PA, Lanko E, Szentesi A, Molnar T, Hagendorn R, Faluhelyi N, Battyani I, Kelemen D, Papp R, Miseta A, Verzar Z, Lerch MM, Neoptolemos JP, Sahin-Toth M, Petersen OH, Hegyi P; Hungarian Pancreatic Study Group. High versus low energy administration in the early phase of acute pancreatitis (GOULASH trial): protocol of a multicentre randomised double-blind clinical trial. BMJ Open. 2017 Sep 14;7(9):e015874. doi: 10.1136/bmjopen-2017-015874. PMID 28912191
- [Background] Parniczky A, Mosztbacher D, Zsoldos F, Toth A, Lasztity N, Hegyi P; Hungarian Pancreatic Study Group and the International Association of Pancreatology. Analysis of Pediatric Pancreatitis (APPLE Trial): Pre-Study Protocol of a Multinational Prospective Clinical Trial. Digestion. 2016;93(2):105-10. doi: 10.1159/000441353. Epub 2015 Nov 26. PMID 26613586
- [Background] Miko A, Eross B, Sarlos P, Hegyi P Jr, Marta K, Pecsi D, Vincze A, Bodis B, Nemes O, Faluhelyi N, Farkas O, Papp R, Kelemen D, Szentesi A, Hegyi E, Papp M, Czako L, Izbeki F, Gajdan L, Novak J, Sahin-Toth M, Lerch MM, Neoptolemos J, Petersen OH, Hegyi P. Observational longitudinal multicentre investigation of acute pancreatitis (GOULASH PLUS): follow-up of the GOULASH study, protocol. BMJ Open. 2019 Sep 3;9(8):e025500. doi: 10.1136/bmjopen-2018-025500. PMID 31481363
- [Background] Zadori N, Gede N, Antal J, Szentesi A, Alizadeh H, Vincze A, Izbeki F, Papp M, Czako L, Varga M, de-Madaria E, Petersen OH, Singh VP, Mayerle J, Faluhelyi N, Miseta A, Reiber I, Hegyi P. EarLy Elimination of Fatty Acids iN hypertriglyceridemia-induced acuTe pancreatitis (ELEFANT trial): Protocol of an open-label, multicenter, adaptive randomized clinical trial. Pancreatology. 2020 Apr;20(3):369-376. doi: 10.1016/j.pan.2019.12.018. Epub 2019 Dec 30. PMID 31959416
- [Background] Parniczky A, Abu-El-Haija M, Husain S, Lowe M, Oracz G, Sahin-Toth M, Szabo FK, Uc A, Wilschanski M, Witt H, Czako L, Grammatikopoulos T, Rasmussen IC, Sutton R, Hegyi P. EPC/HPSG evidence-based guidelines for the management of pediatric pancreatitis. Pancreatology. 2018 Mar;18(2):146-160. doi: 10.1016/j.pan.2018.01.001. Epub 2018 Jan 4. PMID 29398347
- [Background] Hritz I, Czako L, Dubravcsik Z, Farkas G, Kelemen D, Lasztity N, Morvay Z, Olah A, Pap A, Parniczky A, Sahin-Toth M, Szentkereszti Z, Szmola R, Szucs A, Takacs T, Tiszlavicz L, Hegyi P; Magyar Hasnyalmirigy Munkacsoport, Hungarian Pancreatic Study Group. [Acute pancreatitis. Evidence-based practice guidelines, prepared by the Hungarian Pancreatic Study Group]. Orv Hetil. 2015 Feb 15;156(7):244-61. doi: 10.1556/OH.2015.30059. Hungarian. PMID 25661970
- See also: W.H.O. Healthy diet 2018 [Available from: https://www.who.int/news-room/fact-sheets/detail/healthy-diet. — https://www.who.int/news-room/fact-sheets/detail/healthy-diet